CLINICAL TRIAL: NCT07284108
Title: Feasibility, Acceptability, and Preliminary Phase II Efficacy Testing of a Community-Informed Infant Obesity Prevention Program Addressing the Impact of Maternal Mental Health on Eating and Feeding.
Brief Title: Healthy Eating for My Infant: A Community- Informed Infant Obesity Prevention Program Addressing the Impact of Maternal Mental Health on Eating and Feeding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Every Child Succeeds (Unknown)
Responsible Party: Principal Investigator, Cathy Stough, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01DK142998-01 (NIH)
Record Dates: First submitted 2025-11-26; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants randomized into this arm will not receive the study intervention. They will continue to receive standard home visiting services through Every Child Succeeds.
- Intervention (Experimental): Participants randomized into this arm will receive the Healthy Eating for My Infant Intervention (HEMI).
  Interventions: Behavioral: Healthy Eating for My Infant (HEMI)

INTERVENTIONS:
Behavioral: Healthy Eating for My Infant (HEMI) — Our team developed an obesity prevention program, Healthy Eating for My Infant (HEMI), to address the unique factors influencing obesity risk and health behaviors among low-income families and their infants and to be delivered in conjunction with an existing evidence-based home visiting program. HEMI targets healthy feeding with children 3-14 months old through twice monthly behavioral and educational sessions alongside sessions with a peer counselor with similar lived experience to mothers in the program. HEMI incorporates education and evidence-based behavioral techniques (e.g., problem solving, goal setting, behavioral rehearsal) to address topics such as infant nutrition, introduction of solid foods, responsive feeding, realistic healthy eating options, healthy eating on a budget, and recipes). All sessions are delivered in the families' homes. The intervention also includes free grocery delivery and supplemental funds for purchasing foods through grocery delivery.
  Arms: Intervention

SUMMARY:
Infants from low-income families are at increased risk for obesity, but obesity prevention programs tailored specifically to the needs of these infants are lacking. Our team developed Healthy Eating for My Infant (HEMI) to address the specific obesity risk factors, barriers to health behaviors, and needs articulated by community members and low-income families (e.g., maternal mental health, realistic feeding options within the context of food insecurity). The current study will examine the feasibility and acceptability of HEMI delivered via home visiting, as well as preliminary efficacy for improving infant growth trajectories, diet, and parenting/feeding factors related to future obesity risk among infants from low-income families.

ELIGIBILITY:
Inclusion Criteria

* Child age 2 months 0 days to 2 months 30 days at baseline.
* Child is a singleton.
* Mom's must be fluent in English or Spanish.
* Mom must be 18 years or older.

Exclusion Criteria

* Child has major congenital abnormalities or medical conditions requiring specialized feeding.
* Family is currently enrolled in home grocery delivery.

Ages: 2 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Participant Retention | Immediately after the intervention (post-treatment study visit), 6 months after completion of the post-treatment study visit (6 month follow-up visit)
  Participant retention is defined as the percentage of participants that complete each study visit. The percentage of participants completing the post-treatment measurement visit and the 6-month follow-up visit will be calculated, and separate percentages will be calculated for each arm of the study (i.e., control, intervention). This will be measured by tracking yes or no for whether each study visit is completed for each participant.
Treatment Session Completion | Between child age 3 months-14 months (the time period during which the intervention condition is receiving the program).
  The percentage of treatment sessions completed within the designated completion windows will be monitored.
Treatment Acceptability | Between child age 3 months-14 months (the time period during which the intervention condition is receiving the program), Immediately after the intervention (post-treatment study visit)
  Families, peer counselors, and health behavior coaches delivering the program will evaluate program acceptability, utilizing the theoretical framework of acceptability. Families will complete an established questionnaire assessing components of the TFA: affective attitude and effectiveness, coherence and understanding, and perceived burden. The established questionnaire will also be modified to be completed by peer counselors and health behavior coaches to report their perception of acceptability of the program for families. Qualitative interviews will also be conducted with families, peer counselors, and health behavior coaches to identify any modifications to the HEMI program to improve acceptability.
Body Mass Index | Between child ages 3-14 months (when the intervention condition is receiving the program), Immediately after the intervention (post-treatment study visit), 6 months after completion of the post-treatment study visit (6 month follow-up visit).
  Anthropometrics will be measured in triplicate using a calibrated mobile digital SECA baby scale and portable infant length board. Infants will be weighed in a clean diaper without clothes to the nearest 1 gram. The length board has a stable headboard and a moveable foot piece and will be placed on a flat, hard surface. All length measurements will be performed by two team members, with one holding the infant's head straight and flush against the headboard, while the other places one hand across the knees to fully straighten and extend the legs so that heels are at a 90-degree angle against the foot piece and reads the measurement. If holding both legs is not possible, the measurement can be taken with only the right leg extended.
Diet Variety | Immediately after the intervention (post-treatment study visit), 6 months after completion of the post-treatment study visit (6 month follow-up visit).
  Child diet will be assessed via three 24-hour dietary recall interviews conducted with mothers by phone. Trained interviewers, blinded to participant study condition, will employ the USDA automated multiple-pass method, a standardized interview approach demonstrated to improve accuracy of dietary intake data. Data from dietary recalls will be used to calculate diet variety using the minimum dietary diversity (MDD) approach.
Diet Quality | Immediately after the intervention (post-treatment study visit), 6 months after completion of the post-treatment study visit (6 month follow-up visit).
  Child diet will be assessed via three 24-hour dietary recall interviews conducted with mothers by phone. Trained interviewers, blinded to participant study condition, will employ the USDA automated multiple-pass method, a standardized interview approach demonstrated to improve accuracy of dietary intake data. The Nutrition Data Systems for Research (NDSR; Nutrition Coordinating Center, University of Minnesota, Minneapolis, MN) software and foods database will be used to assess total daily energy and macronutrient intake as well as food group servings consumed. Data from dietary recalls will be used to calculate diet quality using the Healthy Eating Index (HEI-Toddlers-2020) for children under age 2 years.
Food Security | Baseline, immediately after the intervention (post-treatment study visit), 6 months after completion of the post-treatment study visit (6 month follow-up visit).
  Food security will be reported using the U.S. Household Food Security Survey Module: Short Form.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
In this proposed project, the raw participant-level data will be shared, along with derived metrics and transformations from initial raw data, with the exception of dietary intake data which will be available after processing by NDSR for nutrient and food servings information. Data will be made available in .csv format or other open file formats and will not require the use of specialized tools to be accessed or manipulated. In accordance with FAIR Principles for data, we will use open file formats (e.g., JPEG, MP4, CSV, TXT, PDF, HTML, etc.) and persistent unique identifiers (PIDs).
Time Frame: Scientific data will be shared as soon as possible. Scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award. The study data will be stored in the repository for at least 5 years.
Access Criteria: All datasets and other information that can be shared will be deposited in UCFigshare, a University of Cincinnati (UC) data repository for NIH-sponsored research at UC. UCFigshare is a platform for accessible and interoperable data sharing and available publicly at https://uc.figshare.com/. Data and other information can be uploaded by NIH-sponsored UC researchers to promote sharing of scientific data in compliance with NIH policy for data management and sharing. UCFigshare provides a data sharing platform consistent with the FAIR (Findability, Accessibility, Interoperability, and Reusability) data principles and is provided via a partnership between the UC Office of Research, UC Libraries, and DTS.

DOCUMENTS (1):
  • Informed Consent Form (2025-11-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT07284108/ICF_000.pdf